CLINICAL TRIAL: NCT01104545
Title: A Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK-3614
Brief Title: A Study of Single Dose MK-3614 (MK-3614-001)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3614-001; MK-3614-001 (Other: Merck); 2010_525
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel A - Healthy (Experimental): Healthy participants receive single oral dose of MK-3614 0.25 mg, 1.25 mg, 0.25 mg w/ food, 0.75 mg or matching placebo. There is at least a 7-day washout between the 4 dosing periods. All doses were administered after an 8-hour fast except for Period 3. Period 3 dose was administered after the ingestion of a high-fat breakfast.
  Interventions: Drug: MK-3614; Drug: Comparator: Placebo
- Panel B - Healthy (Experimental): Healthy participants receive single oral dose of MK-3614 0.5 mg. 0.75 mg, 0.25 mg twice a day (b.i.d.), 0.25 mg three times a day (t.i.d), or matching placebo. There is at least a 7-day washout between the 4 dosing periods. All doses were administered after an 8-hour fast
  Interventions: Drug: MK-3614; Drug: Comparator: Placebo
- Panel C - Hypertensive (Experimental): Hypertensive participants receive single oral dose of MK-3614 0.75 mg. 0.5 mg. 0.75 mg, 0.75 mg or matching placebo. There is at least a 7-day washout between the 4 dosing period. All doses were administered after an 8-hour fast
  Interventions: Drug: MK-3614; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK-3614
Drug: Comparator: Placebo

SUMMARY:
This study will determine if MK-3614, given as single doses, is safe and well tolerated in healthy males and male participants with mild to moderate hypertension.

DETAILED DESCRIPTION:
Up to three planned panels of either 8 healthy participants (Panels A and B) or 8 participants with mild to moderate hypertension (Panel C) will be enrolled. In Panels A and B, 8 participants will alternately receive single rising doses of MK-3614 or placebo. All doses will be administered in the fasted state, except Panel A, Period 3 in which a standard high-fat breakfast provided approximately 30 minutes prior to dosing. Panel A will begin first. At least 3 days will elapse before participants in the alternate panel (Panel B) will receive the next higher dose. In Panel C, 8 mild to moderate hypertensive male participants will receive single rising doses of MK-8892 or placebo. For all panels, there will be at least 7 days washout between treatment periods for any given participant. Participants may only be enrolled in one panel of the study. All participants in periods of all panels (with exception of 0.25 mg fasted/fed periods) will be randomly assigned to either study drug or placebo, i.e., a participant could be assigned to receive study drug in one period and placebo in another. As per the protocol allocation plan, the same participants will receive 0.25 mg MK-3612 in a fasted and fed state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between 18 to 45 years of age; otherwise healthy participants between 18 to 55 years of age newly diagnosed with grade 1 or 2 hypertension
* Participant is in good general health
* Participant is a nonsmoker

Exclusion Criteria:

* Participant has a history of stroke, seizure or major neurological disease
* Participant has functional disability that can interfere with rising from a sitting position to a standing position
* Participant has a family history of a bleeding or clotting disorder
* Participant has a history of cancer
* Participant is unable to refrain from or anticipates the use of any prescription or non-prescription medication during the study
* Participant consumes excessive amounts of alcohol or caffeine
* Participant has had major surgery, donated blood or participated in another investigational study in the past 4 weeks.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2009-05-01 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three panels, each consisting of 8 participants (8 healthy young males in Panel A and Panel B; and 8 with mild-to-moderate hypertension in Panel C) were randomized to receive either MK-3614 or matching placebo in a 3:1 ratio, respectively, in up to 4 treatment periods in Panel A, Panel B and Panel C.
Pre-assignment Details: Each period of each panel (with exception of 0.25 mg fasted/fed periods) will be re-randomized to receive either study drug or placebo, i.e., a participant could be assigned to receive study drug in one period and placebo in another. The same participants will receive 0.25 mg MK-3614 in a fasted and fed state.
Groups:
- Panel A - Healthy: Healthy participants received a single oral dose of MK-3614 0.25 mg, 1.25 mg, 0.25 mg w/ food, 0.75 mg or matching placebo. There was at least a 7-day washout between the 4 dosing periods.
- Panel B - Healthy: Healthy participants received a single oral dose of MK-3614 0.5 mg, 0.75 mg, 0.25 mg twice a day (b.i.d.), 0.25 mg three times a day (t.i.d), or matching placebo. There was at least a 7-day washout between the 4 dosing periods.
- Panel C - Hypertensive: Hypertensive participants received a single oral dose of MK-3614 0.75 mg, 0.5 mg, 0.75 mg, 0.75 mg or matching placebo. There was at least a 7-day washout between the 4 dosing periods.
Period: Overall Study
Arm/Group | Panel A - Healthy | Panel B - Healthy | Panel C - Hypertensive
Started | 8 | 8 | 8 (1 participant received 0.50 mg of MK-3614 or placebo in Periods 3 and 4 instead of planned 0.75 mg)
Completed | 8 | 7 (Participant discontinued after receiving 0.75 mg MK-3614 in Period 1) | 6 (Participants discontinued after receiving MK-3614 0.75 mg (Period 1)and placebo (Period 2))
Not Completed | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A - Healthy | Panel B - Healthy | Panel C - Hypertensive | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (6.8) | 33.4 (7.0) | 46.6 (9.4) | 36.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Reported 1 or More Adverse Event (AE) - Healthy Participants
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants that reported at least 1 AE was summarized. AEs are reported by the dose taken at the time of the event.
Time Frame: up to 7 days for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Groups:
- 0.25 mg MK-3614 Panel A: Participants received a single oral dose of 0.25 mg MK-3614 after an 8-hour fast
- 1.25 mg MK-3614 Panel A: Participants received a single oral dose of 1.25 mg MK-3614 after an 8-hour fast
- 0.25 mg w/ Food MK-3614 Panel A: Participants received a single oral dose of 0.25 mg MK-3614 after ingesting a high-fat breakfest
- 0.75 mg MK-3614 Panel A; 0.75 mg MK-3614 Panel B: Participants received a single oral dose of 0.75 mg MK-3614 after an 8-hour fast
- Placebo Panel A; Placebo Panel B: Participants received a single oral dose of placebo for MK-3614 after an 8-hour fast
- 0.5 mg MK-3614 Panel B: Participants received a single oral dose of 0.50 mg MK-3614 after an 8-hour fast
- 0.25 mg b.i.d. MK-3614 Panel B: Participants received a single daily dose of 0.25 mg MK-3614 b.i.d.
- 0.25 mg t.i.d MK-3614 Panel B: Participants received a single daily oral dose of 0.25 mg MK-3614 t.i.d.
Arm/Group | 0.25 mg MK-3614 Panel A | 1.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A | 0.75 mg MK-3614 Panel A | Placebo Panel A | 0.5 mg MK-3614 Panel B | 0.75 mg MK-3614 Panel B | 0.25 mg b.i.d. MK-3614 Panel B | 0.25 mg t.i.d MK-3614 Panel B | Placebo Panel B
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 7
Percentage of Participants | 100.0 | 100.0 | 80.0 | 33.3 | 66.7 | 66.7 | 66.7 | 20.0 | 60.0 | 57.1

2. Primary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to an AE - Healthy Participants
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants who were discontinued from the study due to an AE were summarized. AEs are reported by the dose taken at the time of the event.
Time Frame: up to 7 days for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | 0.25 mg MK-3614 Panel A | 1.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A | 0.75 mg MK-3614 Panel A | Placebo Panel A | 0.5 mg MK-3614 Panel B | 0.75 mg MK-3614 Panel B | 0.25 mg b.i.d. MK-3614 Panel B | 0.25 mg t.i.d MK-3614 Panel B | Placebo Panel B
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 7
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0

3. Primary Outcome: Percentage of Participants Who Report 1 or More Adverse Event (AE) - Hypertensive Participants
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants that reported at least 1 AE was summarized. The percentage of participants that reported at least 1 AE was summarized. AEs are reported by the dose taken at the time of the event.
Time Frame: up to 7 days for each dose level
Population: All participants in in Panel C who received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Groups:
- 0.75 mg MK-3614 Panel C: Participants received a single oral dose of 0.75 mg MK-3614 after an 8-hour fast
- 0.5 mg MK-3614 Panel C: Participants received a single oral dose of 0.5 mg MK-3614 after an 8-hour fast
- Placebo Panel C: Participants received a single oral dose of placebo for MK-3614 after an 8-hour fast
Arm/Group | 0.75 mg MK-3614 Panel C | 0.5 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 8 | 5 | 7
Percentage of Participants | 75.0 | 60.0 | 57.1

4. Primary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to an AE - Hypertensive Participants
Description: as for outcome 2
Time Frame: up to 7 days for each dose level
Population: All participants in in Panel C who received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | 0.75 mg MK-3614 Panel C | 0.5 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 8 | 5 | 7
Percentage of Participants | 12.5 | 0.0 | 14.3

5. Primary Outcome: Area Under the Concentration Time-curve From Hour 0 to Infinity (AUC0-inf) of MK-3614 - Healthy Participants
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the AUC0-inf of MK-3614 in healthy participants.
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and who complied with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: nM•h
Arm/Group | 0.25 mg MK-3614 Panel A | 1.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A | 0.75 mg MK-3614 Panel A | 0.5 mg MK-3614 Panel B | 0.75 mg MK-3614 Panel B | 0.25 mg b.i.d. MK-3614 Panel B | 0.25 mg t.i.d MK-3614 Panel B
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 6 | 6 | 5 | 5
nM•h | 83.8 (53.1) | 412.0 (96.4) | 83.8 (9.46) | 223.0 (83.1) | 173.0 (82.0) | 168.0 (27.7) | NA (NA) — AUC0-inf not calculated for multiple dose arms | NA (NA) — AUC0-inf not calculated for multiple dose arms

6. Primary Outcome: Maximum Concentration (Cmax) of MK-3614- Healthy Participants
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the Cmax of MK-3614 in healthy participants.
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | 0.25 mg MK-3614 Panel A | 1.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A | 0.75 mg MK-3614 Panel A | 0.5 mg MK-3614 Panel B | 0.75 mg MK-3614 Panel B | 0.25 mg b.i.d. MK-3614 Panel B | 0.25 mg t.i.d MK-3614 Panel B
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 5 | 5
nM | 4.9 (1.68) | 29.8 (5.20) | 3.6 (1.09) | 17.0 (4.48) | 11.5 (4.22) | 13.4 (2.24) | 5.1 (0.55) | 7.1 (1.50)

7. Primary Outcome: Time to Cmax (Tmax) of MK-3614- Healthy Participants
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the Tmax of MK-3614 in healthy participants.
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: as for outcome 5
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | 0.25 mg MK-3614 Panel A | 1.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A | 0.75 mg MK-3614 Panel A | 0.5 mg MK-3614 Panel B | 0.75 mg MK-3614 Panel B | 0.25 mg b.i.d. MK-3614 Panel B | 0.25 mg t.i.d MK-3614 Panel B
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 5 | 5
hour (hr) | 4.0 [4.0 to 12.0] | 4.0 [2.0 to 6.0] | 6.0 [6.0 to 6.0] | 4.0 [4.0 to 6.0] | 4.0 [4.0 to 8.0] | 4.0 [2.0 to 6.0] | 4.0 [4.0 to 4.0] | 16.0 [16.0 to 18.0]

8. Primary Outcome: Apparent Terminal Half-life (t1/2) of MK-3614- Healthy Participants
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the t1/2 of MK-3614 in healthy participants.
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | 0.25 mg MK-3614 Panel A | 1.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A | 0.75 mg MK-3614 Panel A | 0.5 mg MK-3614 Panel B | 0.75 mg MK-3614 Panel B | 0.25 mg b.i.d. MK-3614 Panel B | 0.25 mg t.i.d MK-3614 Panel B
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 5 | 5
hr | 9.2 (4.5) | 10.1 (2.3) | 13.1 (1.2) | 9.1 (3.0) | 9.7 (3.6) | 9.5 (2.1) | 11.7 (4.1) | 14.7 (6.0)

9. Primary Outcome: Area Under the Concentration Time-curve From Hour 0 to Infinity (AUC0-inf) of MK-3614 - Hypertensive Participants
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the AUC0-inf of MK-3614 in hypertensive participants
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: All participants in in Panel C who received at least 1 dose of study drug and who complied with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model and had available data for the endpoint. Data were summarized by dose taken and not by sequence.
Measure: Mean (Standard Deviation); unit: nM•h
Arm/Group | 0.75 mg MK-3614 Panel C | 0.5 mg MK-3614 Panel C
Number analyzed (Participants) | 8 | 5
nM•h | 253.0 (52.0) | 134.0 (39.5)

10. Primary Outcome: Maximum Concentration (Cmax) of MK-3614- Hypertensive Participants
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the Cmax of MK-3614 in hypertensive participants
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | 0.75 mg MK-3614 Panel C | 0.5 mg MK-3614 Panel C
Number analyzed (Participants) | 8 | 5
nM | 19.1 (3.88) | 10.9 (1.55)

11. Primary Outcome: Time to Cmax (Tmax) of MK-3614- Hypertensive Participants
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the Tmax of MK-3614 in hypertensive participants
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | 0.75 mg MK-3614 Panel C | 0.5 mg MK-3614 Panel C
Number analyzed (Participants) | 8 | 5
hr | 4.0 [2.0 to 4.0] | 4.0 [4.0 to 4.0]

12. Primary Outcome: Apparent Terminal Half-life (t1/2) of MK-3614 of MK-3614- Hypertensive Participants
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the t1/2 of MK-3614 in hypertensive participants
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | 0.75 mg MK-3614 Panel C | 0.5 mg MK-3614 Panel C
Number analyzed (Participants) | 8 | 5
hr | 9.1 (2.8) | 8.7 (1.4)

13. Primary Outcome: Change From Baseline in Heart Rate - Healthy Participants
Description: Heart rate measurements were obtained using a validated, semi-automated oscillometric device. The difference between the predose (baseline) measurement and the measurement 24 obtained 24 hours postdose was summarized. Data for each specific dose were combined regardless of panel.
Time Frame: Baseline and 24 hours post-dose for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Groups:
- 0.25 mg MK-3614: Participants received single oral dose of 0.25 mg MK-3614 either after an 8 -hour fast or after a high-fat breakfast.
- 0.25 mg Twice a Day (b.i.d.) MK-3614: Participants received single daily dose of 0.25 mg MK-3614 b.i.d.
- 0.25 mg t.i.d MK-3614: Participants received single daily oral dose of 0.25 mg MK-3614 t.i.d.
- 0.5 mg MK-3614: Participants received a single oral dose of 0.50 mg MK-3614 after an 8-hour fast
- 0.75 mg MK-3614: Participants received a single oral dose of 0.75 mg MK-3614 after an 8-hour fast
- 1.25 mg MK-3614: Participants received a single daily dose of 1.25 mg MK-3614
- Placebo: Participants received a single oral dose of placebo for MK-3614 after an 8-hour fast
Arm/Group | 0.25 mg MK-3614 | 0.25 mg Twice a Day (b.i.d.) MK-3614 | 0.25 mg t.i.d MK-3614 | 0.5 mg MK-3614 | 0.75 mg MK-3614 | 1.25 mg MK-3614 | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 12 | 6 | 13
Beats per minute (bpm) | -4.7 (3.7) | -0.6 (7.2) | 5.4 (7.2) | 2.5 (4.8) | -0.3 (5.9) | 6.3 (11.8) | 3.8 (6.6)

14. Primary Outcome: Change From Baseline in Brachial Arterial Systolic Blood Pressure - Healthy Participants
Description: Brachial arterial systolic blood pressure measurements were obtained using a validated, semi-automated oscillometric device. The difference between the predose (baseline) measurement and the measurement 24 obtained 24 hours postdose was summarized. Data for each specific dose were combined regardless of panel.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.25 mg MK-3614 | 0.25 mg Twice a Day (b.i.d.) MK-3614 | 0.25 mg t.i.d MK-3614 | 0.5 mg MK-3614 | 0.75 mg MK-3614 | 1.25 mg MK-3614 | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 12 | 6 | 13
mmHg | -3.3 (4.8) | 2.4 (2.3) | -2.6 (5.3) | -1.0 (9.2) | -3.1 (5.7) | -3.0 (8.0) | -0.2 (7.4)

15. Primary Outcome: Change From Baseline in Brachial Arterial Diastolic Blood Pressure - Healthy Participants
Description: Brachial arterial diastolic blood pressure measurements were obtained using a validated, semi-automated oscillometric device. The difference between the predose (baseline) measurement and the measurement 24 obtained 24 hours postdose was summarized. Data for each specific dose were combined regardless of panel.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.25 mg MK-3614 | 0.25 mg Twice a Day (b.i.d.) MK-3614 | 0.25 mg t.i.d MK-3614 | 0.5 mg MK-3614 | 0.75 mg MK-3614 | 1.25 mg MK-3614 | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 12 | 6 | 13
mmHg | -1.7 (3.1) | 0.8 (6.7) | -2.8 (5.4) | -1.0 (5.6) | -1.8 (4.0) | 3.2 (6.0) | -0.6 (3.3)

16. Primary Outcome: Change From Baseline in Heart Rate - Hypertensive Participants
Description: HR measurements were obtained using a validated, semi-automated oscillometric device. The difference between the predose (baseline) measurement and the measurement 24 obtained 24 hours postdose was summarized. Data for each specific dose were combined regardless of sequence.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in in Panel C who received at least 1 dose of study drug and who complied with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- 0.5 mg MK-3614 Panel C: Participants received a single oral dose of 0.50 mg MK-3614 after an 8-hour fast
Arm/Group | 0.5 mg MK-3614 Panel C | 0.75 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 5 | 8 | 7
bpm | 0.7 (8.1) | 0.8 (10.7) | -8.4 (8.5)

17. Primary Outcome: Change From Baseline in Brachial Arterial Systolic Blood Pressure - Hypertensive Participants
Description: Brachial arterial systolic blood pressure measurements were obtained using a validated, semi-automated oscillometric device. The difference between the predose (baseline) measurement and the measurement 24 obtained 24 hours postdose was summarized. Data for each specific dose were combined regardless of sequence.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.5 mg MK-3614 Panel C | 0.75 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 5 | 8 | 7
mmHg | -5.2 (14.2) | -10.0 (13.0) | -18.1 (15.6)

18. Primary Outcome: Change From Baseline in Brachial Arterial Diastolic Blood Pressure - Hypertensive Participants
Description: Brachial arterial diastolic blood pressure measurements were obtained using a validated, semi-automated oscillometric device. The difference between the predose (baseline) measurement and the measurement 24 obtained 24 hours postdose was summarized. Data for each specific dose were combined regardless of sequnce.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- 0.5 mg MK-3614 Panel C: Participant received single oral dose of 0.5 mg of MK-3614 after an 8 -hour fast
Arm/Group | 0.5 mg MK-3614 Panel C | 0.75 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 5 | 8 | 7
mmHg | 0.3 (9.3) | -4.4 (6.5) | -9.1 (6.9)

19. Secondary Outcome: Area Under the Concentration Time-curve From Hour 0 to Infinity (AUC0-inf) of 0.25 mg MK-3614 - Healthy Participants- Fasted Versus Fed
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the AUC0-inf of 0.25 mg MK-3614 in healthy participant when administered after an 8 hour fast and after a high-fat breakfest.
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: All participants in Panels A who received at least 1 dose of study drug and who complied with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: nM•h
Arm/Group | 0.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A
Number analyzed (Participants) | 6 | 4
nM•h | 83.8 (53.1) | 83.8 (9.46)
Statistical Analysis 1: Comparison: 0.25 mg MK-3614 Panel A vs 0.25 mg w/ Food MK-3614 Panel A; Test type: Other; Geometric mean ratio (GMR) = 1.0 — GMR = Fed/Fasted

20. Secondary Outcome: Maximum Concentration (Cmax) of 0.25 mg MK-3614 - Healthy Participants- Fasted Versus Fed
Description: Blood samples taken at Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose of each dosing period to determine the Cmax of 0.25 mg MK-3614 when administered after an 8 hour fast and after a high-fat breakfest.
Time Frame: Predose, and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose for each dose level
Population: All participants in Panel A who received at least 1 dose of study drug and who complied with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | 0.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A
Number analyzed (Participants) | 6 | 5
nM | 4.85 (1.68) | 3.56 (1.09)
Statistical Analysis 1: Comparison: 0.25 mg MK-3614 Panel A vs 0.25 mg w/ Food MK-3614 Panel A; Test type: Other; GMR = 0.73 — GMR = Fed/fasted

21. Secondary Outcome: Percentage Change From Baseline in Augmentation Index (AIx) at 24 Hours Postdose - Healthy Participants
Description: Augmentation index was measured at predose (baseline), and 1, 4, 8, 12, and 24 hours postdose by aplanation tonometry of radial artery. The change from baseline at 24 hours postdose was summarized. Data for each specific dose were combined regardless of panel.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- 0.25 mg b.i.d. MK-3614: Participants received single daily dose of 0.25 mg MK-3614 b.i.d.
Arm/Group | 0.25 mg MK-3614 | 0.25 mg b.i.d. MK-3614 | 0.25 mg t.i.d MK-3614 | 0.5 mg MK-3614 | 0.75 mg MK-3614 | 1.25 mg MK-3614 | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 12 | 6 | 13
Percentage change | -4.7 (10.1) | -5.2 (7.9) | -0.8 (3.1) | -1.8 (6.0) | -3.0 (4.0) | -1.5 (6.0) | 0.8 (4.1)

22. Secondary Outcome: Percentage Change From Baseline in Augmentation Index (AIx) at 24 Hours Postdose - Hypertensive Participants
Description: Augmentation index was measured at predose (baseline), and 1, 4, 8, 12, and 24 hours postdose by aplanation tonometry of radial artery. The change from baseline at 24 hours postdose was summarized.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panel C who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 0.5 mg MK-3614 Panel C | 0.75 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 5 | 8 | 7
Percentage change | 2.0 (6.4) | -2.3 (4.9) | 1.1 (5.0)

23. Secondary Outcome: Percentage Change From Baseline in Bleeding Time at 24 Hours Postdose - Healthy Participants
Description: Blood was to be drawn at predose (baseline) and 3 and 24 hours postdose and bleeding time was to be assessed using a Newborn Surgicutt device. Change in bleeding time from baseline at 24 hours postdose were to be summarized. Due to change in number of blood draws and total blood volume restrictions, bleeding time assessment was not performed as planned.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Arm/Group | 0.25 mg MK-3614 | 0.25 mg b.i.d. MK-3614 | 0.25 mg t.i.d MK-3614 | 0.5 mg MK-3614 | 0.75 mg MK-3614 | 1.25 mg MK-3614 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Percentage Change From Baseline in Bleeding Time at 24 Hours Postdose- Hypertension Participants
Description: as for outcome 23
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panel C who received at least 1 dose of study drug and had available data for endpoint.
Arm/Group | 0.5 mg MK-3614 Panel C | 0.75 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Percentage Change in Cyclic Guanosine Monophosphate (GMP) From Baseline at 24 Hours Postdose - Healthy Participants
Description: Blood was drawn at predose (baseline) and 1, 4, 8, and 24 hours postdose. The change in cyclic GMP at 24 hours postdose was summarized. Due to change in number of blood draws and total blood volume restrictions, data for GMP were only collected for first 2 periods of each panel. Therefore only limited data were available and summarized. Data for each specific dose were combined regardless of panel.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 0.25 mg MK-3614 | 0.25 mg b.i.d. MK-3614 | 0.25 mg t.i.d MK-3614 | 0.5 mg MK-3614 | 0.75 mg MK-3614 | 1.25 mg MK-3614 | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 0 | 12 | 6 | 11
Percentage change | 0.1 (0.1) | 0.0 (0.0) | 0.2 (0.1) |  | 0.0 (0.1) | 0.0 (0.0) | 0.0 (0.1)

26. Secondary Outcome: Percentage Change in Cyclic Guanosine Monophosphate (GMP) From Baseline at 24 Hours Postdose - Hypertension Participants
Description: Blood was drawn at predose (baseline) and 1, 4, 8, and 24 hours postdose. The change in cyclic GMP at 24 hours postdose was summarized. Due to change in number of blood draws and total blood volume restrictions, data for GMP were only collected for first 2 periods of each panel. Therefore only limited data were available and summarized.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panel C who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 0.5 mg MK-3614 Panel C | 0.75 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 0 | 6 | 2
Percentage change |  | 0.2 (0.2) | 0.0 (0.2)

27. Secondary Outcome: Percentage Change From Baseline in Platelet Aggregation at 24 Hours Postdose - Healthy Participants
Description: Platelet aggregation induced by adenosine diphosphate (ADP) was measured at predose (baseline) and 3 and 24 hours postdose. Percent inhibition from baseline at 24 hours postdose was calculated. Due to change in number of blood draws and total blood volume restrictions, data for platelet aggregation were only collected for first 2 periods of each panel. Therefore only limited data were available and summarized. Data for each specific dose were combined regardless of panel.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panels A and B who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 0.25 mg MK-3614 | 0.25 mg b.i.d. MK-3614 | 0.25 mg t.i.d MK-3614 | 0.5 mg MK-3614 | 0.75 mg MK-3614 | 1.25 mg MK-3614 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 0 | 3
Percentage change |  |  |  |  | -22.3 (26.3) |  | -5.0 (12.8)

28. Secondary Outcome: Percentage Change From Baseline in Platelet Aggregation at 24 Hours Postdose - Hypertensive Participants
Description: Platelet aggregation induced by adenosine diphosphate (ADP) was measured at predose (baseline) and 3 and 24 hours postdose. Percent inhibition from baseline at 24 hours postdose was calculated. Due to change in number of blood draws and total blood volume restrictions, data for platelet aggregation were only collected for first 2 periods of each panel. Therefore only limited data were available and summarized.
Time Frame: Baseline and 24 hours postdose for each dose level
Population: All participants in Panel C who received at least 1 dose of study drug and had available data for endpoint.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 0.5 mg MK-3614 Panel C | 0.75 mg MK-3614 Panel C | Placebo Panel C
Number analyzed (Participants) | 0 | 6 | 2
Percentage change |  | -9.3 (12.9) | -19.5 (21.9)

ADVERSE EVENTS:
Time Frame: Up to 7 days postdose for each dose level (up to 15 weeks total)
Description: All participants that received at least 1 dose of study drug and had data available for endpoint.
Groups:
- 0.75 mg MK-3614 Panel A; 0.75 mg MK-3614 Panel C: Participant received a single oral dose of 0.75 mg MK-3614 after an 8-hour fast
- Placebo Panel C: Participant received a single oral dose of placebo for MK-3614 after an 8-hour fast
Arm/Group | 0.25 mg MK-3614 Panel A | 1.25 mg MK-3614 Panel A | 0.25 mg w/ Food MK-3614 Panel A | 0.75 mg MK-3614 Panel A | Placebo Panel A | 0.5 mg MK-3614 Panel B | 0.75 mg MK-3614 Panel B | 0.25 mg b.i.d. MK-3614 Panel B | 0.25 mg t.i.d MK-3614 Panel B | Placebo Panel B | 0.75 mg MK-3614 Panel C | 0.5 mg MK-3614 Panel C | Placebo Panel C
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/7 | 0/8 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/7 | 0/8 | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/5 | 2/6 | 4/6 | 4/6 | 4/6 | 1/5 | 3/5 | 4/7 | 6/8 | 3/5 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.25 mg MK-3614 Panel A (N=6) | 1.25 mg MK-3614 Panel A (N=6) | 0.25 mg w/ Food MK-3614 Panel A (N=5) | 0.75 mg MK-3614 Panel A (N=6) | Placebo Panel A (N=6) | 0.5 mg MK-3614 Panel B (N=6) | 0.75 mg MK-3614 Panel B (N=6) | 0.25 mg b.i.d. MK-3614 Panel B (N=5) | 0.25 mg t.i.d MK-3614 Panel B (N=5) | Placebo Panel B (N=7) | 0.75 mg MK-3614 Panel C (N=8) | 0.5 mg MK-3614 Panel C (N=5) | Placebo Panel C (N=7)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood immunoglobulin E increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure orthostatic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (24) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (21) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic heart rate response increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysstasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 3 (6) | 1 (2) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vibratory sense increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.